CLINICAL TRIAL: NCT06864741
Title: Acute Stroke Rehabilitation Using a Low-cost Virtual Reality Platform: a Pilot Study.
Brief Title: Virtual Reality Rehabilitation for Stroke Patients in the Hospital and at Home.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Acadia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 70851
Record Dates: First submitted 2025-02-26; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Stroke Acute
Keywords: stroke; rehabilitation; motor disorder; virtual reality
MeSH Terms: conditions — Stroke; Motor Disorders

STUDY DESIGN:
Intervention Model Description: During the in-hospital phase, the study model is a parallel design. During the at-home phase, the study model is a crossover design. Participants may enroll in one or both phases of the study.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- In Hospital - Standard of Care (No Intervention): Inpatient standard of care for acute stroke
- In Hospital - Virtual Reality Rehabilitation (Experimental): Inpatient supplementary rehabilitation delivered through a virtual reality headset
  Interventions: Behavioral: Virtual reality guided motor rehabilitation
- At Home - Standard of care (No Intervention): Outpatient standard of care for acute stroke
- At Home - Virtual Reality Rehabilitation (Experimental): Outpatient supplementary rehabilitation delivered through a virtual reality headset
  Interventions: Behavioral: Virtual reality guided motor rehabilitation

INTERVENTIONS:
Behavioral: Virtual reality guided motor rehabilitation — Custom rehabilitation exercises running on a Meta Quest 2/3S/3 head mounted virtual reality display.
  Arms: At Home - Virtual Reality Rehabilitation; In Hospital - Virtual Reality Rehabilitation

SUMMARY:
The goal of this clinical trial is to test whether a low-cost virtual reality (VR) motor rehabilitation platform can improve motor recovery in people recovering from a first-time ischemic stroke both in the hospital and at home. The study focuses on adults aged 18 and older who have experienced moderate to severe upper limb motor deficits.

The main questions it aims to answer are:

* Can VR-based motor therapy improve upper limb motor function compared to standard care?
* Is VR-based motor therapy a feasible and acceptable treatment option for stroke patients?

Researchers will compare patients receiving VR therapy to those receiving standard care to see if the VR therapy leads to greater improvements in motor recovery and more positive patient experiences.

Participants will:

* Complete standardized assessments of motor function and quality of life at multiple time points.
* Participate in VR therapy sessions (if in the treatment group), using gamified activities designed to improve upper limb movement.
* Provide feedback on their experience with the VR system, including ease of use, motion sickness, and engagement.

This study will help determine whether VR-based rehabilitation can be a practical, effective way to improve access to therapy and recovery outcomes for stroke patients, especially in rural settings with limited rehabilitation resources.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of first-time ischemic stroke involving the middle cerebral artery, confirmed by CT or MRI;
* score between 6 and 40 on Fugl-Meyer Assessment's Upper Limb Extremity Subscore (FM - UE), indicating moderate to severe motor deficit;
* ability and willingness to provide consent (score of 18 or more on the Montreal Cognitive Assessment) or assent (for scores lower than 18 on MoCA with consent provided by an authorized third party with the necessary legal authority to consent on behalf of patient)
* INPATIENT ARM: less than 5 weeks since stroke onset with admission to Valley Regional Hospital in Kentville, NS, Canada
* OUTPATIENT ARM: less than 3 months since stroke onset with discharge to home setting located within 1 hour drive of Valley Regional Hospital in Kentville, NS, Canada

Exclusion Criteria:

* brainstem, cerebellar or bilateral stroke lesion
* a secondary neurological condition (e.g., Parkinson's disease)
* musculoskeletal injuries interfering with task performance
* an uncorrected visual deficit due to stroke or other etiologies
* apraxia as identified by clinical assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Treatment effectiveness in hospital | From enrollment to one week following the end of treatment at day 26
  Measure if patients receiving supplementary VR motor therapy show improved motor recovery compared to receiving standard care in hospital using the Fugl-Meyer Assessment's Upper Limb Extremity Subscore. Values range from 0 to 66 with lower scores indicating a larger motor deficit.
Treatment effectiveness at home | From enrollment through standard of care and VR treatment completion on Day 47
  Measure if patients receiving supplementary VR motor therapy show improved motor recovery compared to receiving standard care for home-based patients using the Fugl-Meyer Assessment's Upper Limb Extremity Subscore. Values range from 0 to 100 with lower scores indicating a larger motor deficit.
Treatment feasibility - Motion Sickness | From enrollment to one week following the end of treatment
  Measure motion sickness levels immediately after each therapy sessions using the Virtual Reality Sickness Questionnaire. Values range from 0 to 100 with higher scores indicating more reported motion sickness.
Treatment feasibility - Attitudes towards technology | From enrollment to one week following the end of treatment
  Measure attitudes towards the VR technology before and after the intervention using a VR Attitudes Survey. Values range from 0 to 6 with higher scores indicating more favorable attitudes towards the VR technology.
Patient engagement at home | From enrollment through standard of care and VR treatment completion on Day 47
  Assess patient engagement with adaptive at-home rehabilitation using the percentage of daily sessions completed. Values range from 0% to 100% with higher scores indicating a higher rate of session completion.

SECONDARY OUTCOMES:
Treatment effectiveness - Motor performance | From enrollment to one week following the end of treatment
  Measure if patients receiving VR motor therapy show improved motor performance using the Box and Blocks Test. Values range from 0 to 150 with higher scores indicating improved motor performance.
Treatment effectiveness - Quality of life | From enrollment to one week following the end of treatment
  Measure if patients receiving VR motor therapy show reduced disability and improved health-related quality of life using the Stroke Impact Scale. Values range from 0 to 100 with higher scores indicating reduced disability and higher quality of life.
VR motor assessment validity | From enrollment to one week following the end of treatment
  Examine the validity of a VR motor assessment for monitoring stroke motor recovery trajectories in the real world. This will be explored by comparing data between the real-world and virtual Box and Blocks tests which will result in a correlation coefficient ranging from 0 to 1 with a higher value indicating a stronger alignment in metrics.
Gender differences in acceptance of VR rehabilitation technology | From enrollment to one week following the end of treatment
  Analyze differences between women and men in relation to the acceptance of VR treatment, using the VR Attitudes Survey. Values range from 0 to 6 with higher scores indicating more favorable attitudes towards the VR technology.
Independent use of home-based VR treatment | From enrollment through standard of care and VR treatment completion on Day 47
  By meeting certain criteria during the study, participants can qualify to complete VR sessions on their own. Measure the proportion of participants qualifying for independent operation.
Performance characteristics of stroke patients | From enrollment to last VR rehabilitation session
  Measure motor performance for each task over time using motor performance z-scores. Mean scores equal zero with deviations indicating distance in standard deviations from the mean (with no minimum or maximum). Higher scores indicate better motor performance.
Barriers to treatment adoption | From enrollment to one week following the last VR session
  Qualitative feedback will be analyzed thematically to identify potential barriers and enablers of adopting VR stroke rehabilitation. This qualitative analysis does not use a quantitative scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Valley Regional Hospital, Kentville, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Given the small sample size and single recruitment site, the investigators are uncertain if confidentiality can be ensured with sharing IPD. The investigators will address this with the institution's Research Ethics Board.